CLINICAL TRIAL: NCT04435665
Title: A Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Phase 2a Study to Determine Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Activity of NFX-179 Gel in Subjects With Cutaneous Neurofibromas
Brief Title: NFX-179 Topical Gel Treatment in Adults With Neurofibromatosis 1 (NF1) and Cutaneous Neurofibromas (cNF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NFlection Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NFX-179-NF1-201
Record Dates: First submitted 2020-06-08; First posted 2020-06-17 (Actual); Results first posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-07

CONDITIONS: Neurofibromatosis 1; Cutaneous Neurofibroma
Keywords: NFX-179
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NFX-179 Gel Low (Experimental): NFX-179 Gel for topical administration, once daily for 28 days
  Interventions: Drug: NFX-179 Gel
- NFX-179 Gel Mid (Experimental): NFX-179 Gel for topical administration, once daily for 28 days
  Interventions: Drug: NFX-179 Gel
- NFX-179 Gel High (Experimental): NFX-179 Gel for topical administration, once daily for 28 days
  Interventions: Drug: NFX-179 Gel
- Vehicle Arm (Placebo Comparator): Vehicle Gel, for topical administration, once daily for 28 days
  Interventions: Drug: Vehicle Gel

INTERVENTIONS:
Drug: NFX-179 Gel — gel for topical administration
  Arms: NFX-179 Gel High; NFX-179 Gel Low; NFX-179 Gel Mid
Drug: Vehicle Gel — vehicle gel for topical administration
  Arms: Vehicle Arm

SUMMARY:
This study will enroll and treat subjects with cutaneous neurofibromas with NFX-179, a topical study drug. Eligible subjects will receive treatment for 28 days and be observed by a study doctor for approximately 56 days. Subjects will be randomly assigned to 1 of 4 treatment groups. 3 of the treatment groups will receive a specific dose NFX-179, and 1 group will receive placebo. The subject, study doctor, and NFlection Therapeutics will not know what treatment group each subject is assigned. Study participation requires at least 7 clinic visits, blood, urine, and tissue collection, images of the treated cutaneous neurofibromas, electrocardiograms, and information regarding the subject's medical and disease history.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age
2. Subject must provide written informed consent prior to any study procedures
3. Subject must have a clinical diagnosis of NF1
4. Subject has 6 Study cNF Tumors (5 Target cNF Tumors [1 on the face; 4 on the anterior trunk or upper extremities] that will be treated with the assigned study medication;1 Untreated cNF Tumor on the anterior trunk or upper extremities) that each meet the following criteria:

   * Has, in the investigator's opinion, a clinically typical appearance
   * Is dome shaped
   * Is not pedunculated
   * Is a discrete tumor
   * Is not irritated
   * Is not in an area subject to repeated trauma (e.g., area that is shaved, on the beltline, under a bra strap, etc.)
   * Does not have an active cutaneous infection
   * Has a diameter that is ≥5mm and ≤10mm
   * Has a height of ≥2mm
   * Is, when centered in the center of the provided template, the only cNF tumor visible
   * Is not within 5mm of the orbital rim.
5. Subject is willing to have the 5 Target cNF Tumors and the 1 Untreated cNF Tumor excised at the end of the treatment period
6. Subject is willing to have hair in the area surrounding the Target cNF Tumors shaved, if necessary, to obtain photographs
7. Subject is willing to minimize exposure of each Target cNF to natural and artificial ultraviolet radiation
8. Subject is willing to forego treatment of the Target cNF Tumors, except protocol specified therapy, during the study
9. Female subjects who are women of childbearing potential must have a negative urine pregnancy test result and be willing to use a protocol approved, contraceptive method for the duration of the study
10. Subject is willing and able to follow all study instructions and to attend all study visits.

Exclusion Criteria:

1. Subject has applied any of the following topical products in the previous 30 days on or in proximity to any Study cNF Tumor that, in the investigator's opinion, impairs evaluation of any the tumor or which exposes the subject to an unacceptable risk by study participation:

   * Corticosteroids
   * Retinoids (e.g., tazarotene, tretinoin, adapalene)
   * > 5% of an alpha-hydroxy acid (e.g., glycolic acid, lactic acid)
   * Fluorouracil
   * Imiquimod
2. Any Study cNF Tumor has ever been treated with an MEK inhibitor or a BRAF inhibitor
3. The subject has used any of the following systemic medications in the noted time period:

   * Retinoids (e.g., etretinate, isotretinoin) within the previous 90 days
   * MEK inhibitors within the previous 180 days
   * BRAF inhibitors within the previous 180 days
4. Subject has a history of hypersensitivity to any of the ingredients in the study medications
5. Subject has any known intercurrent illness or physical condition that would, in the investigator's opinion, impair evaluation of a Target cNF Tumor or which exposes the subject to an unacceptable risk by study participation
6. Subject has, in the investigator's opinion, clinically relevant history of liver disease, including viral hepatitis, current alcohol abuse, or cirrhosis
7. Subject has a history of metastatic disease, or active cancer (excluding nonmelanoma skin cancer, Stage I cervical cancer, ductal carcinoma in situ of the breast, or Stage 0 chronic lymphocytic lymphoma) within the previous 5 years
8. Subject has any condition (e.g., other skin conditions or diseases, metabolic dysfunction, physical examination findings, clinical laboratory findings) or situation (e.g., vacation, scheduled surgery) that would, in the investigator's opinion, impair evaluation of a Target cNF Tumor or which exposes the subject to an unacceptable risk by study participation
9. Subject has participated in an investigational drug trial in which administration of an investigational study medication occurred within the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Webster, MD, PhD, Study Director — NFlection Therapeutics
Locations (6):
- United States (6):
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Skin Search of Rochester, Inc., Rochester, New York
  - DermResearch, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The Education & Research Foundation, Inc., Lynchburg, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- NFX-179 Gel Low (0.05%): NFX-179 Gel for topical administration, once daily for 28 days
  NFX-179 Gel 0.05%
  NFX-179 Gel: gel for topical administration
- NFX-179 Gel Mid (0.15%): NFX-179 Gel for topical administration, once daily for 28 days
  NFX-179 Gel 0.15%
  NFX-179 Gel: gel for topical administration
- NFX-179 Gel High (0.50%): NFX-179 Gel for topical administration, once daily for 28 days
  NFX-179 Gel 0.50%
  NFX-179 Gel: gel for topical administration
- Vehicle Arm (Placebo): Vehicle Gel, for topical administration, once daily for 28 days
  Vehicle Gel placebo
  Vehicle Gel: vehicle gel for topical administration
Period: Overall Study
Arm/Group | NFX-179 Gel Low (0.05%) | NFX-179 Gel Mid (0.15%) | NFX-179 Gel High (0.50%) | Vehicle Arm (Placebo)
Started | 12 | 11 | 12 | 13
Completed | 12 | 11 | 12 | 12
Not Completed | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NFX-179 Gel Low (0.05%) | NFX-179 Gel Mid (0.15%) | NFX-179 Gel High (0.50%) | Vehicle Arm (Placebo) | Total
Number analyzed (Participants) | 12 | 11 | 12 | 13 | 48
Age, Continuous [Mean (Full Range); unit: years] | 51.1 [31 to 69] | 49.5 [29 to 73] | 43.5 [25 to 63] | 45.2 [33 to 72] | 47.8 [25 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 8 | 7 | 32
  Male | 3 | 3 | 4 | 6 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-white | 1 | 4 | 2 | 2 | 9
  White | 11 | 7 | 10 | 11 | 39
  Asian | 0 | 3 | 0 | 1 | 4
  Black/African American | 1 | 1 | 2 | 1 | 5
  Hispanic or Latino | 2 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 9 | 7 | 9 | 11 | 36
  Not reported | 1 | 4 | 2 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Phospho-erk (p-ERK) Levels of Target cNF Tumors in NFX-179 Gel Group and Vehicle Gel Group After 28 Days of Once-daily (QD) Application
Description: Pharmacodynamic activity (biochemical and physiologic effects of drugs) of NFX-179 Gel as defined by suppression of phospho-ERK (p-ERK) levels in Target cNF Tumors in each NFX-179 Gel group compared with the Vehicle Gel group after 28 days of once-daily (QD) application will be measured at Week 4
Time Frame: Baseline through Week 4
Population: The p-ERK analysis included all available p-ERK data from tumors determined by histology to be cNF tumors. Missing data were due to missing or non-analyzable tumor samples or tumor samples shown to come from non-cNF tumors upon histologic review. Therefore the number of participants is not the same as those in the participant flow.
Measure: Mean (Standard Deviation); unit: % reduction in pERK to total ERK
Units Other Than Participants: Tumors
Arm/Group | Vehicle Arm (Placebo) | NFX-179 Gel Low (0.05%) | NFX-179 Gel Mid (0.15%) | NFX-179 Gel High (0.50%)
Number analyzed (Participants) | 12 | 11 | 10 | 11
Number analyzed (Tumors) | 53 | 53 | 47 | 53
% reduction in pERK to total ERK | 0.3054 (0.1369) | 0.2734 (0.1257) | 0.2267 (0.1272) | 0.1627 (0.0686)

2. Primary Outcome: Safety and Tolerability of NFX-179 Gel Measured by Local Tolerability Assessment
Description: Safety and tolerability will be measured via a local tolerability assessment. The investigator will assess erythema, edema, scabbing/crusting, vesiculation, and erosion. The subject will assess stinging, burning, and pruritus. All assessments are performed using a 4-point scale (0 none, 1 mild, 2 moderate, 3 severe).
Time Frame: Baseline through Week 4
Measure: Number; unit: events
Arm/Group | Vehicle Arm (Placebo) | NFX-179 Gel Low (0.05%) | NFX-179 Gel Mid (0.15%) | NFX-179 Gel High (0.50%)
Number analyzed (Participants) | 13 | 12 | 11 | 12
events
  subject reported instances of mild pruritus | 2 | 5 | 7 | 4
  subject reported instances of moderate pruritus | 0 | 1 | 2 | 0
  subject reported instances of mild burning | 6 | 0 | 0 | 0
  subject reported instances of mild stinging | 0 | 0 | 0 | 4
  investigator reported instances of mild erythema | 0 | 2 | 1 | 1
  investigator reported instances of moderate erythema | 0 | 0 | 0 | 1
  investigator reported instances of mild edema | 0 | 0 | 1 | 0
  investigator reported instances of scabbing/crusting | 0 | 0 | 0 | 1

3. Primary Outcome: Assessment of Adverse Events
Description: Assessment of adverse events (AEs)
Time Frame: Baseline through Week 8
Measure: Number; unit: Subjects
Arm/Group | Vehicle Arm (Placebo) | NFX-179 Gel Low (0.05%) | NFX-179 Gel Mid (0.15%) | NFX-179 Gel High (0.50%)
Number analyzed (Participants) | 13 | 12 | 11 | 12
Subjects
  Number of subjects with treatment-emergent AEs | 2 | 2 | 1 | 3
  Number of subects with related treatment-emergent AEs | 0 | 0 | 0 | 1
  Number of subjects withdrawn due to AEs | 0 | 0 | 0 | 0
  Subjects with mild treatment-emergent AEs | 1 | 0 | 0 | 3
  Subjects with moderate treatment-emergent AEs | 1 | 2 | 1 | 0
  Subjects with severe treatment-emergent AEs | 0 | 0 | 0 | 0

4. Secondary Outcome: Percent Change in cNF Tumor Volume (Cubic Millimeters)
Description: Percent change in cNF tumor volume after 28 days of QD applications of NFX-179 gel based on tumor volume derived from ruler measurements.
Time Frame: Baseline through Week 4
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Vehicle Arm (Placebo) | NFX-179 Gel Low (0.05%) | NFX-179 Gel Mid (0.15%) | NFX-179 Gel High (0.50%)
Number analyzed (Participants) | 13 | 12 | 11 | 12
percentage change | -8.0 (18.2) | -1.6 (22.1) | -11.9 (29.4) | -16.7 (30.3)

5. Secondary Outcome: Systemic Exposure of NFX-179 Gel Measured by Plasma Concentration
Description: Systemic exposure of NFX-179 will be measured during the 28 days of QD applications at select investigative sites. Pharmacokinetic samples will be drawn at the baseline visit and week 4 visit. 5 time point samples will be collected at the week 4 visit.
Time Frame: Baseline through Week 4
Population: Pharmacokinetic data from subjects treated with active NFX-179 gel was performed, which does not include samples from subjects treated with Vehicle gel (placebo). As such, no analysis pharmacokinetic analysis was performed in the Vehicle Arm.
Measure: Number; unit: ng/mL
Arm/Group | Vehicle Arm (Placebo) | NFX-179 Gel Low (0.05%) | NFX-179 Gel Mid (0.15%) | NFX-179 Gel High (0.50%)
Number analyzed (Participants) | 0 | 1 | 2 | 1
ng/mL
  Baseline, pre dose (0 hour) |  | NA — below the lower limit of quantification | NA — below the lower limit of quantification | NA — below the lower limit of quantification
  Week 4, pre dose (0 hour) |  | NA — below the lower limit of quantification | NA — below the lower limit of quantification | 0.439
  Week 4, post dose 30 min |  | NA — below the lower limit of quantification | NA — below the lower limit of quantification | 0.887
  Week 4, post dose 1 hour |  | NA — below the lower limit of quantification | NA — below the lower limit of quantification | 0.573
  Week 4, post dose 2 hours |  | NA — below the lower limit of quantification | NA — below the lower limit of quantification | 0.718
  Week 4, post dose 4 hours |  | NA — below the lower limit of quantification | NA — below the lower limit of quantification | 0.528

6. Secondary Outcome: Change in Physician Assessment of Tumor Severity Score
Description: Effect of treatment with The Physician Tumor Assessment is the investigator's assessment of the average overall severity of each Target cNF tumor at a particular time point. The Physician Tumor Assessment is a 5-point measuring tumor severity (0 clear/none, 1 almost clear, 2 mild, 3 moderate, 4 severe). The assessment is performed at the Baseline visit and week 4 visit.
Time Frame: Baseline through Week 4
Measure: Mean (Standard Deviation); unit: Change in Investigator Assessment score
Arm/Group | Vehicle Arm (Placebo) | NFX-179 Gel Low (0.05%) | NFX-179 Gel Mid (0.15%) | NFX-179 Gel High (0.50%)
Number analyzed (Participants) | 12 | 12 | 11 | 12
Change in Investigator Assessment score
  Visit 2 | 2.74 (0.53) | 2.46 (0.62) | 2.60 (0.57) | 2.65 (0.70)
  Visit 5 | 2.51 (0.58) | 3.58 (0.62) | 2.50 (0.59) | 2.70 (0.67)

7. Secondary Outcome: Change in Subject Self-Assessment of Tumor Severity Score
Description: The Subject Self-Assessment is the subject's assessment of the average overall severity of each Target cNF at a particular time point and is not a comparison with any other time point. The Subject Self-Assessment is a 5-point measuring tumor severity (0 clear/none, 1 almost clear, 2 mild, 3 moderate, 4 severe). The assessment is performed at the Baseline visit and week 4 visit.
Time Frame: Baseline through Week 4
Measure: Mean (Standard Deviation); unit: change in subject assessment score
Arm/Group | Vehicle Arm (Placebo) | NFX-179 Gel Low (0.05%) | NFX-179 Gel Mid (0.15%) | NFX-179 Gel High (0.50%)
Number analyzed (Participants) | 12 | 12 | 11 | 12
change in subject assessment score
  Visit 2 | 2.75 (0.73) | 2.81 (0.53) | 2.71 (0.38) | 2.38 (0.71)
  Visit 5 | 2.50 (0.60) | 2.76 (0.55) | 2.50 (0.56) | 2.39 (0.61)

ADVERSE EVENTS:
Time Frame: Up to 56 Days
Arm/Group | Vehicle Arm (Placebo) | NFX-179 Gel Low (0.05%) | NFX-179 Gel Mid (0.15%) | NFX-179 Gel High (0.50%)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 2/13 | 2/12 | 2/11 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Arm (Placebo) (N=13) | NFX-179 Gel Low (0.05%) (N=12) | NFX-179 Gel Mid (0.15%) (N=11) | NFX-179 Gel High (0.50%) (N=12)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple allergies (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corona test positive (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menopause (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (5):
  • Study Protocol and Statistical Analysis Plan: Full Protocol (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT04435665/Prot_SAP_000.pdf
  • Study Protocol: Amendment 1 (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT04435665/Prot_001.pdf
  • Study Protocol: Amendment 2 (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/65/NCT04435665/Prot_002.pdf
  • Study Protocol: Amendment 3 (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT04435665/Prot_003.pdf
  • Informed Consent Form (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/65/NCT04435665/ICF_004.pdf